CLINICAL TRIAL: NCT07256405
Title: Contribution of Metagenomic Sequencing Using Nanopore Technology to the Management of Post-traumatic Bone and Joint Infections
Brief Title: Metagenomic Next-Generation Sequencing for the Diagnosis of Fracture-related Infection
Acronym: METADIAG 2
Status: Active, not recruiting | Type: Observational
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Collaborators: Military Teaching Hospital Sainte Anne, Toulon (Unknown); Institut Hospitalo-Universitaire Méditerranée Infection (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-CHITS-017
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Infection; Fracture; Bone
Keywords: Nanopore; Fracture; Metagenomic; Trauma; Infection; High throughput sequencing
MeSH Terms: conditions — Infections; Fractures, Bone; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tissue samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fracture-related infection: Patients suspected of having acute or chronic post-traumatic osteoarticular infection according to the criteria of the FRI (Fracture-Related Infection) consensus group and scheduled to undergo a bone and/or soft tissue biopsy as part of routine care
  Interventions: Diagnostic Test: Metagenomic sequencing

INTERVENTIONS:
Diagnostic Test: Metagenomic sequencing — Samples shall be submitted to high throughput sequencing using both illumine MiSeq and Oxford Nanopore Technologies.

SUMMARY:
The value of next-generation sequencing (NGS) using Nanopore technology has been demonstrated in the case of diabetic patients' wounds or in prosthetic joint infections. The aim of this study is to demonstrate its relevance as a new diagnostic approach for fracture-related infections (FRI).

Bone samples from patient with FRI will be submitted to shotgun metagenomic Next-generation sequencing using Oxford Nanopore Technology (ONT) in order to establish its diagnostic value in this context in comparison with the reference method.

DETAILED DESCRIPTION:
Tissue samples from patients with FRI used for routine culture and remaining after this step will be retrieved for metagenomic sequencing.

Both DNA extraction and host-DNA depletion steps will be performed. The nanopore ligation sequencing protocol along with native barcoding will be used to carry out DNA library preparation. Sequencing will be run using ONT GridION device. The generated reads will be computerized to be assigned at each taxonomic levels. The results will be compared to those of routine diagnosis to determine NGS concordance with culture.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of fracture-related infection (FRI consensus group)
* Patient scheduled to undergo a bone and/or soft-tissue biopsy as part of routine care

Exclusion Criteria:

* Patient opposition
* Patient under a legal protection measure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to hospital following trauma for whom a fracture-related infection was diagnosed.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2024-03-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Concordance between the microbiological documentation obtained by sequencing and that of the reference technique (culture) | 1 month
  Metagenomic sequencing will be used to determine the microbiome of fracture-related infections.
  Data will be compared with those of reference microbiological identification techniques (culture).

SECONDARY OUTCOMES:
Time to obtain final microbiological results by sequencing compared with the reference technique (culture) | 1 month
  Duration (in days) for definitive microbiological diagnosis using both culture and NGS-based protocols.
Number of cases in which an adjustment of targeted antibiotic therapy would be made based on NGS results. | 1 month
  Number of cases in which an adjustment of targeted antibiotic therapy would be made based on NGS results.
Microbial abundance defined by the number of reads (sequence reads) obtained per phylotype | 1 month
  To describe the microbiome of fracture related infection in terms of microbial diversity and abundance in order to discuss both raw reads number and relative abundance roles when considering NGS results in this context.

CONTACTS AND LOCATIONS:
Overall Officials: LACÔTE-DELARBRE David, MD, Study Director — Military Teaching Hospital Sainte Anne
Locations (2):
- France (2):
  - IHU, service des maladies infectieuses chroniques, Marseille, Bouches-du-Rhône
  - Military Teaching Hospital Sainte Anne, Toulon, VAR

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tarabichi M, Shohat N, Goswami K, Alvand A, Silibovsky R, Belden K, Parvizi J. Diagnosis of Periprosthetic Joint Infection: The Potential of Next-Generation Sequencing. J Bone Joint Surg Am. 2018 Jan 17;100(2):147-154. doi: 10.2106/JBJS.17.00434. PMID 29342065
- [Result] Goswami K, Shope AJ, Tokarev V, Wright JR, Unverdorben LV, Ly T, Chen See J, McLimans CJ, Wong HT, Lock L, Clarkson S, Parvizi J, Lamendella R. Comparative meta-omics for identifying pathogens associated with prosthetic joint infection. Sci Rep. 2021 Dec 9;11(1):23749. doi: 10.1038/s41598-021-02505-7. PMID 34887434
- [Result] Sanderson ND, Street TL, Foster D, Swann J, Atkins BL, Brent AJ, McNally MA, Oakley S, Taylor A, Peto TEA, Crook DW, Eyre DW. Real-time analysis of nanopore-based metagenomic sequencing from infected orthopaedic devices. BMC Genomics. 2018 Sep 27;19(1):714. doi: 10.1186/s12864-018-5094-y. PMID 30261842
- [Result] Ivy MI, Thoendel MJ, Jeraldo PR, Greenwood-Quaintance KE, Hanssen AD, Abdel MP, Chia N, Yao JZ, Tande AJ, Mandrekar JN, Patel R. Direct Detection and Identification of Prosthetic Joint Infection Pathogens in Synovial Fluid by Metagenomic Shotgun Sequencing. J Clin Microbiol. 2018 Aug 27;56(9):e00402-18. doi: 10.1128/JCM.00402-18. Print 2018 Sep. PMID 29848568
- [Result] Walter N, Orbenes N, Rupp M, Alt V. The State of Research in Fracture-Related Infection-A Bibliometric Analysis. Medicina (Kaunas). 2022 Aug 29;58(9):1170. doi: 10.3390/medicina58091170. PMID 36143847